CLINICAL TRIAL: NCT03534440
Title: Assessment of Left Ventricle Diastolic Function in High Risk Patients Undergoing Major Vascular Surgery as an Early Indicator of Cardiac Failure. Observational Study
Brief Title: Assessment of Diastolic Function in High Risk Patients Undergoing Major Vascular Surgery
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mateusz Zawadka, Principal Investigator, Medical University of Warsaw
Other Study IDs: DD-TEVAR-2018
Record Dates: First submitted 2018-04-15; First posted 2018-05-23 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Diastolic Dysfunction; Heart Failure; Aneurysm Aortic
Keywords: Diastolic Dysfunction; Anesthesia; Preoperative assessment; Postoperative care; TEVAR
MeSH Terms: conditions — Heart Failure; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients scheduled for Thoracic Endovascular Aortic Repair (TEVAR) surgery will have transthoracic echocardiography evaluation of left ventricle diastolic function during the perioperative period.

DETAILED DESCRIPTION:
Patients undergoing TEVAR surgery are a high risk group of developing perioperative cardiovascular complications.

Left ventricle diastolic dysfunction is common in this group of patients because of the prevalence of risk factors: > 60 years old, hypertension, smoking history and diabetes.

Because of many predisposing factors that occur during the surgery: stress respond, fluid shifts, anaesthesia and mechanical ventilation. Deterioration of the diastolic function is likely to occur in perioperative period

In this study, the investigators will evaluate change in left ventricle diastolic function as a marker for early detection of a myocardial failure in patients scheduled for an elective TEVAR surgery. The examination will be performed preoperatively, shortly after the surgery and 24 hours after the surgery.

Aim: The aim of the study is to evaluate the diastolic function of left ventricle in perioperative period after high risk surgery. This may provide a valuable information in preoperative risk stratification and postoperative therapy guidance.

ELIGIBILITY:
Inclusion Criteria:

* scheduled TEVAR
* >60 years old

Exclusion Criteria:

* Atrial fibrillation or other non-sinus rhythms
* Atrioventricular blocks
* Heart rate change more than 25% postoperatively
* Not adequate transthoracic view
* Postoperative shock
* Sepsis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a Thoracic Endovascular Aortic Repair
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in left ventricle diastolic function in time | Baseline, 2 hours and 24 hours
  Echocardiographic assessment of change in left ventricle diastolic function repeated in time intervals:
  Baseline before the surgery, 2 and 24 hours after the surgery

SECONDARY OUTCOMES:
Change in biochemistry markers: troponins | Baseline, 2 hours and 24 hours
  Assessment of change in level of troponins. Baseline before the surgery, 2 and 24 hours after the surgery
Change in biochemistry markers: brain natriuretic peptide | Baseline, 2 hours and 24 hours
  Assessment of change in level of brain natriuretic peptide. Baseline before the surgery, 2 and 24 hours after the surgery
Change in left ventricle systolic function | Baseline, 2 hours and 24 hours
  Echocardiographic assessment of change in left ventricle systolic function repeated in time intervals:
  Baseline before the surgery, 2 and 24 hours after the surgery
Hemodynamic parameters: Heart rate | Baseline, 2 hours and 24 hours
  Heart rate during echocardiography evaluation.
Hemodynamic parameters: Systolic and diastolic pressure | Baseline, 2 hours and 24 hours
  Systolic and diastolic pressure measurements during echocardiography evaluation. Record vasopressors requirement.
Fluid balance | 72 hours
  Monitoring of diuresis hourly, fluid losses and fluids intake
Kidney function | 72 hours
  Monitoring of glomerular filtration rate and requirement for a dialysis daily
Length of stay in hospital | up to 14 days
  Documentation of length of stay in hospital since the surgery
Mortality | up to 30 days
  Documentation of in-hospital mortality and 30 days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Of Warsaw, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: Undecided